CLINICAL TRIAL: NCT06680726
Title: Research Collaboration for a Precision Oncology Program (POP)
Acronym: POP
Status: Recruiting | Type: Observational
Sponsor: Andreas Wicki (Other)
Collaborators: Hoffmann-La Roche (Industry); University of Zurich (Other); University Hospital, Zürich (Other)
Responsible Party: Sponsor-Investigator, Andreas Wicki, Professor, University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: POP; 2022-02289 (Other: Kantonale Ethikkommission Zürich (KEK Zürich))
Record Dates: First submitted 2024-10-30; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Cancer
Keywords: cancer; real world data (RWD); clinical decision-making; precision oncology; advanced diagnostics; tumor tissue imaging
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Matching with RWD — A set of clinical and genetic data are matched to generate a RWD cohort for comparison.
Other: Imaging Mass Cytometry — Protein expression patterns in tumor tissue and tumor microenvironment are analyzed by Imaging Mass Cytometry.

SUMMARY:
The Precision Oncology Program (POP) research collaboration aims to help generate information about the individual tumour biology for patients with advanced malignancies, using innovative biotechnologies and patient profile comparison ("matching") against specific databases (Real-world data, RWD) and to inform about potential benefit, or lack of benefit, from a given treatment.

DETAILED DESCRIPTION:
This is an observational clinical project. The aim of this research collaboration is to establish processes to advance precision oncology within the clinical routine. POP generates information about individual tumour for patients with advanced cancers using innovative molecular technologies and patient profile comparison ("matching") against specific public and non-public databases with the aim to support clinical decision-making (therapy prediction).

The POP report will summarize the clinically-relevant findings from the following tests and procedures:

A. Routine genetic testing:

FMI (routine genetic testing) Comprehensive tumour genotyping which includes alterations in cancer-relevant genes and the following parameters: Tumor mutational burden (TMB), Loss of heterozygosity (LoH), Microsatellite Instability (MSI).

B. POP-specific additional testing:

1. Research grade: Imaging Mass Cytometry (IMC) To better capture tumour heterogeneity beyond genetics, and to inform therapy decisions of whether or not a particular treatment may show efficacy, we will perform IMC on existing formalin-fixed paraffin-embedded (FFPE) tissue sections. IMC technology enables quantification of over 40 selected proteins and protein modifications, while simultaneously interrogating phenotype and cell signaling. It allows identification of markers predictive of response (or resistance) of individual cancer patients, and enables the analysis of tumour tissues at single-cell resolution, capturing characteristics of the tumour cells, the tumour microenvironments and the relationship between tumour, stromal and immune compartments. The analysis of the tumour at the protein level and the spatial distribution of the different compartments will significantly increase and broaden the routine genetic analysis to identify potentially druggable alterations.
2. Patient Matching Against Cancer Databases The patient matching will be performed by Roche using the Flatiron Health-Foundation Medicine Clinico-genomic Database (FH-FMI CGDB).

The following scenarios will be explored as part of the project:

(i) a comparison of clinical data (e.g. entity, TNM classification, previous therapies, etc) to extract similar clinical phenotypes and the related treatment history and outcomes (clinical level) (ii) a comparison at the genotype level (genomic level) (iii) a combination of the possibilities above.

The POP report will be shared with the Molecular Tumour Board (MTB) and discussed in the absence of the treating physician. The MTB will consider all available information at its own discretion and in adherence to the available standard guidelines. However, only treatment recommendations based on routine diagnostics will be forwarded to the treating physician. Hypothetical MTB's treatment decisions based on the POP summary report will not be forwarded the treating physician.

NOTE: All additional project specific recommendations remain non-prescriptive and will not be forwarded to the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* In the case of deceased persons: signed general consent
* All patients with the diagnosis of a solid tumour including adenocarcinoma, squamous cell carcinoma, neuroendocrine carcinoma, sarcoma, etc
* ECOG-performance status 0-2, if applicable
* Willing and able to understand all project related procedures, including transfer of coded (i.e. pseudonymised) or anonymized clinical data to external partners (e.g. Roche), if applicable

Exclusion Criteria:

* Patients with the diagnosis of blood cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with histology based proven diagnosis of cancer; all stages and subtypes can be included. Pre-cancerous lesions, e.g. DCIS, LCIS, CIN, etc. cannot be included.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Utility of RWD matching report as assessed by the questionnaire | From date of enrollment, assessed up to 2 years
  1. Is the Report used to identify imminent or future treatment options?
  2. How has the Report changed your confidence in the primary decision?
  3. Does the Report support the primary therapy decision?
  4. Is the relevant information in the Report non supportive of the Resources used or the primary therapy decision?
  5. What Resources did you use for the primary therapy decision?
  6. How useful was the Report to decide on the secondary therapy decision?
  7. Which features of the Report were used for the secondary therapy decision?
  8. Could you have gathered the information in the Report used for the secondary treatment decision in less than 15 min?
  9. Did the Report provide unique information on personalizing future treatment regimens?
Utility of the IMC report as assessed by the questionnaire | From date of enrollment, assessed up to 2 years
  1. Is the Report used to identify imminent or future treatment options?
  2. How has the Report changed your confidence in the primary decision?
  3. Does the Report support the primary therapy decision?
  4. Is the relevant information in the Report non supportive of the Resources used or the primary therapy decision?
  5. What Resources did you use for the primary therapy decision?
  6. How useful was the Report to decide on the secondary therapy decision?
  7. Which features of the Report were used for the secondary therapy decision?
  8. Could you have gathered the information in the Report used for the secondary treatment decision in less than 15 min?
  9. Did the Report provide unique information on personalizing future treatment regimens?

SECONDARY OUTCOMES:
Number of POP reports provided | through study completion, an average of 1 year
  Number (proportion) of patients in which the POP reports could be provided to the MTB
Classification of Treatment Options | through study completion, an average of 1 year
  Type of treatment recommendations made by the MTB

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zürich (Universitätsspital Zürich), Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boos LA, Doerig C, Gut G, Miglino N, Fabregas Ibanez L, Rizzo S, Scharfe Fruechtenicht C, Chitale N, Lu C, Zoche M, Bodenmiller B, Chevrier S, Eklund AS, Nowak M, Rahmani Khajouei S, Berardo CG, Kaczmarek L, Bosshard K, Archey W, Bodmer M, Glinz D, Camarillo-Retamosa E, Hempel CL, Rahimzadeh P, Gosztonyi B, Richter U, Bankel L, Wicki A. Precision Oncology Program (POP), an observational study using real-world data and imaging mass cytometry to explore decision support for the Molecular Tumor Board: study protocol. BMJ Open. 2025 Mar 26;15(3):e096591. doi: 10.1136/bmjopen-2024-096591. PMID 40139698